CLINICAL TRIAL: NCT06159647
Title: Consumer Responses to Alcohol Warnings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anna Grummon, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 71682
Record Dates: First submitted 2023-11-27; First posted 2023-12-07 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Larynx, Artificial; Drugs, Generic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alcohol Messages (Experimental): Participants view 12 messages: 10 messages related to health topics (2 messages for each of 5 randomly selected health topics from among all health topics) and 2 control messages.
  Interventions: Behavioral: Mouth cancer warning; Behavioral: Throat cancer warning; Behavioral: Voice box (larynx) warning; Behavioral: Esophagus cancer warning; Behavioral: Liver cancer warning; Behavioral: Colon and rectum cancer warning; Behavioral: Breast cancer; Behavioral: Cancer (generic, not site-specific); Behavioral: Addiction and neurological changes; Behavioral: Hypertension; Behavioral: Liver damage; Behavioral: Harm to fetus; Behavioral: Dementia; Behavioral: Impaired sleep; Behavioral: Drinking guidelines; Behavioral: Control; Behavioral: Road injuries

INTERVENTIONS:
Behavioral: Mouth cancer warning — Participants will view messages about the risk of mouth cancer from alcohol consumption.
Behavioral: Throat cancer warning — Participants will view messages about the risk of throat cancer from alcohol consumption.
Behavioral: Voice box (larynx) warning — Participants will view messages about the risk of voice box (larynx) cancer from alcohol consumption.
Behavioral: Esophagus cancer warning — Participants will view messages about the risk of esophagus cancer from alcohol consumption.
Behavioral: Liver cancer warning — Participants will view messages about the risk of liver cancer from alcohol consumption.
Behavioral: Colon and rectum cancer warning — Participants will view messages about the risk of colon and rectum cancer from alcohol consumption.
Behavioral: Breast cancer — Participants will view messages about the risk of breast cancer from alcohol consumption.
Behavioral: Cancer (generic, not site-specific) — Participants will view messages about the risk of cancer (not site-specific) from alcohol consumption.
Behavioral: Addiction and neurological changes — Participants will view messages about the risk of addiction and neurological changes from alcohol consumption.
Behavioral: Hypertension — Participants will view messages about the risk of hypertension from alcohol consumption.
Behavioral: Liver damage — Participants will view messages about the risk of liver damage from alcohol consumption.
Behavioral: Harm to fetus — Participants will view messages about the risk of harm to a fetus from alcohol consumption during pregnancy.
Behavioral: Dementia — Participants will view messages about the risk of dementia from alcohol consumption.
Behavioral: Impaired sleep — Participants will view messages about the risk of impaired sleep from alcohol consumption.
Behavioral: Drinking guidelines — Participants will view messages about guidelines for alcohol consumption.
Behavioral: Control — Participants will view neutral messages unrelated to the harms of alcohol consumption.
Behavioral: Road injuries — Participants will view messages about the risk of road injuries from alcohol consumption.

SUMMARY:
The primary objective is to evaluate whether alcohol warnings about different topics elicit higher perceived message effectiveness than control messages. The secondary objective is to evaluate whether alcohol warnings about different topics elicit higher reactance than control messages.

DETAILED DESCRIPTION:
Participants will complete a within-subjects online randomized experiment in which they will view and rate messages on the risk of alcohol consumption. Participants will view and rate 12 messages total: 10 warning messages and 2 control messages. They will rate each message on perceived message effectiveness (primary outcome) and message reactance (secondary outcome). The 10 warning messages will be about 5 different warning topics (i.e., 2 messages per topic) and the 2 control messages will be about 1 control topic (2 messages per topic). In this within-subjects experiment, the survey will present the topics in random order and the messages within each topic in random order.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and older
* Reside in the United States
* Able to complete a survey in English

Exclusion Criteria:

* Under 21 years of age
* Reside outside the United States
* Unable to complete a survey in English

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2522 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Perceived message effectiveness | The survey will take up to 20 minutes.
  The study will assess perceived message effectiveness using 1 item: "How much does this message discourage you from wanting to drink alcohol?" Response options will range from "not at all" (coded as 1) to "a great deal" (coded as 5). Higher scores indicate more perceived message effectiveness.

SECONDARY OUTCOMES:
Reactance | The survey will take up to 20 minutes.
  The study will assess reactance using 1 item: "Say how much you disagree or agree with this statement: This message exaggerates the health effects of alcohol." Response options will range from "strongly disagree" (coded as 1) to "strongly agree" (coded as 5). Higher scores indicate more reactance.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Grummon, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Online study, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will post de-identified individual participant data in a publicly available repository.
Supporting Information: SAP, Analytic Code
Time Frame: Investigators will post IDP upon acceptance of any manuscripts associated with the data generated in this study.
Access Criteria: Data and code will be publicly available.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/47/NCT06159647/Prot_SAP_000.pdf